CLINICAL TRIAL: NCT06416189
Title: The Decrowding Rate Post Premolar Extraction With and Without Fixed Appliance: Randomized Controlled Trial
Brief Title: Teeth Decrowding With and Without Fixed Appliances
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Samer Mheissen (Other)
Responsible Party: Principal Investigator, Samer Mheissen, Researcher, Samer Mheissen
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Ortho-0001
Record Dates: First submitted 2024-01-26; First posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Tooth Crowding
MeSH Terms: conditions — Malocclusion | interventions — Orthodontic Appliances, Fixed

STUDY DESIGN:
Intervention Model Description: Two groups; one with fixed braces and one without fixed braces.
Who Masked: Participant, Outcomes Assessor
Masking Description: The two groups will have lingual arches. However, patients without braces will not be informed about their braces before 5 months of trial initiation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Braces (Active Comparator): Fixed appliance would be bonded post teeth extraction (premolars). subsequently, leveling and alignment using sequence of archwires would be followed. The measurements would be done using models each month.
  Interventions: Device: Fixed appliances
- Without braces (No Intervention): Extraction of premolars and only observing the case over time. The measurements would be done using models each month.

INTERVENTIONS:
Device: Fixed appliances — MBT Brackets 0.022 inch
  Arms: Braces

SUMMARY:
In orthodontics, the teeth tend to move to the extraction space. This tooth movement becomes of larger importance when there is a crowding. During the COVID lockdown period, It was noted that some cases have a significant improvement and almost all the crowding was relieved without appliance activation.

DETAILED DESCRIPTION:
In this randomized controlled trial, a sufficient number of patients would be randomly assigned into two groups; one with braces and one without fixed braces.

ELIGIBILITY:
Inclusion Criteria:

- Patients with permanent dentition between age group of 13 - 30 years.

* Maxillary or mandibular crowding >4.1mm and requiring extraction of maxillary first premolars or mandibular first premolars. The crowding will be measured using a caliper one cast models.
* Fully erupted teeth from 1st molar to the 1st molar.
* Patients with periodontally sound dentition.
* Patients with good general health. No previous history of extraction or orthodontic tooth movement.

Exclusion Criteria:

* Cases requiring orthognathic surgery.

  * History of systemic and medical illness.
  * Contraindication of extraction.
  * Previous history of orthodontic treatment.
  * Poor oral hygiene.
  * Nickel allergy.

Ages: 13 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-02-02 (Actual); Primary Completion 2024-08-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Anterior teeth alignment every 4 weeks at each time point. | 6 months
  The cumulative before extraction and space closure for 4 months (mean difference before and after)..

SECONDARY OUTCOMES:
Molar anchorage loss at each time point. | 6 months
  The anchorage loss of molars will be measured over time using the models.
Gingival invagination | 9 months
  this will be measured by visual inspection intraorally.

CONTACTS AND LOCATIONS:
Overall Officials: Samer Mheissen, DDS, Principal Investigator — Private Practice
Locations (1):
- Medical Services, Amman, Jordan

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP
Time Frame: 12 months